CLINICAL TRIAL: NCT06648330
Title: The Effect of Blood Lactate Levels on Postoperative Gastrointestinal Morbidity After Paraaortic Retroperitoneal Lymph Node Dissection
Brief Title: Blood Lactate Level With Paraaortic Lymph Node Dissection
Status: Completed | Type: Observational
Sponsor: Duygu Akyol (Other Government)
Responsible Party: Sponsor-Investigator, Duygu Akyol, Principal investigator, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Organization: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Other Study IDs: 2023-544
Record Dates: First submitted 2024-09-23; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-05

CONDITIONS: Morbidity; Gynaecologic Cancer
Keywords: major open gynaecological cancer surgery; paraaortic lymph node dissection; gastrointestinal complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gynaecological cancer surgeries with paraaortic retroperitoneal lymph node dissection: Paraaortic retroperitoneal lymph node dissection was performed in 75 patients with gynaecological cancer surgery
  Interventions: Procedure: Paraaortic retroperitoneal lymph node dissection

INTERVENTIONS:
Procedure: Paraaortic retroperitoneal lymph node dissection — The relationship between lactate level and mesenteric ischaemia in gynaecological cancer surgeries with paraaortic retroperitoneal lymph node dissection will be evaluated.

SUMMARY:
This study was designed as a prospective observational study.

DETAILED DESCRIPTION:
In this study, the investigator planned to evaluate the effect of blood lactate levels on postoperative gastrointestinal morbidity after paraaortic retroperitoneal lymph node dissection. In gynaecological surgeries, following the removal of the intestines from the surgical field, the retroperitoneal space is entered and the main vessels such as the vena cava inferior and aorta are accessed through the left or right approach depending on the experience and habit of the per-operative surgeon, and total systemic lymph node dissection or bulky lymph node excision is performed depending on the case. During the removal of the intestines from the surgical field, hypoperfusion may develop due to decreased blood flow to the intestines. for this purpose, the investigator planned to investigate the relationship between the change in blood gas lactate values and postoperative gastrointestinal complications in this process.

ELIGIBILITY:
Inclusion Criteria:

* 18 years

  * Patients undergoing paraaortic retroperitoneal lymph node dissection

Exclusion Criteria:

* Patients with chronic lung disease
* Patients with inflammatory bowel disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Gynaecological cancer surgeries with paraaortic retroperitoneal lymph node dissection
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
intraoperative lactate levels | intraoperatively
  Change from baseline in lactate levels in paraaortic lymph node dissection

CONTACTS AND LOCATIONS:
Locations (1):
- Duygu, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mothes H, Wickel J, Sponholz C, Lehmann T, Kaluza M, Zanow J, Doenst T. Monitoring of the Progression of the Perioperative Serum Lactate Concentration Improves the Accuracy of the Prediction of Acute Mesenteric Ischemia Development After Cardiovascular Surgery. J Cardiothorac Vasc Anesth. 2021 Jun;35(6):1792-1799. doi: 10.1053/j.jvca.2021.02.007. Epub 2021 Feb 8. PMID 33663981
- [Result] Oh TK, Song IA, Jeon YT. Peri-operative serum lactate level and postoperative 90-day mortality in a surgical ICU: A retrospective association study. Eur J Anaesthesiol. 2020 Jan;37(1):31-37. doi: 10.1097/EJA.0000000000001117. PMID 31724965
- [Result] Selcuk I, Oz M, Toyran A, Tatar I, Engin-Ustun Y, Demiryurek D. Para-aortic lymphadenectomy: step by step surgical education video. J Turk Ger Gynecol Assoc. 2021 Aug 31;22(3):253-254. doi: 10.4274/jtgga.galenos.2019.2019.0117. Epub 2019 Aug 9. PMID 31397548